CLINICAL TRIAL: NCT04595721
Title: Comparison of Physical Versus Visual Distraction in the Reduction of Pain During Local Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resident did not have sufficient time to start study before graduating and leaving institution
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20020881
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Pain
Keywords: Dental pain
MeSH Terms: conditions — Pain; Toothache

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (No Intervention): Participants will receive standard injection procedures
- Visual distraction (Active Comparator): Participants engage in visual distraction during the injection procedures
  Interventions: Behavioral: Hidden object
- Physical distraction (Active Comparator): Participants engage in physical distraction during the injection procedures
  Interventions: Behavioral: Stress ball

INTERVENTIONS:
Behavioral: Hidden object — Participant will be instructed to look at the hidden object image on the overhead light to look for a number of objects and observe the image.
  Arms: Visual distraction
Behavioral: Stress ball — Participants will be handed a single-use, squeezable stress ball and instructed to squeeze the stress ball.
  Arms: Physical distraction

SUMMARY:
The purpose of this study is to compare physical versus visual distractions to determine which technique reduces perceived pain better during local anesthesia injections.

DETAILED DESCRIPTION:
Before the local anesthesia injection, patients will be asked to give a preliminary VAS score based on what level of pain 0-10 they anticipate they will feel during the local anesthesia injection. Following the injection the participant will be asked to quantify the pain felt during the injection on a 0-10 Visual analog scale (VAS). The VAS scores will only be taken from the first injection of the appointment. Participants will be asked their gender, race, age, geographic location they spent most of their lives as well. Participants will be de-identified and randomly assigned a number that will be recorded along with their collected data on a two-factor, password protected web server. Information collected during this study may be used for further analysis and publication.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing a dental procedure that requires a buccal infiltration with Septocaine 1:100,000 epinephrine (EPI) (Articaine hydrochloride 4% and EPI 1:100,000) or an inferior alveolar nerve block injection with 2% lidocaine with 1:100,000 epinephrine.
* Adults greater than 18 years old.
* Patients with limited English proficiency will be included only if their primary language is Spanish.

Exclusion Criteria:

* Patients with a known or suspected allergy to anesthetic agent, sulfites, amide-type local anesthetic, or to any ingredient in anesthetic solutions will not be included.
* Any patients taking medications affecting pain response on the day of the dental appointment.
* Children younger than 18 years old.
* Patients with limited English proficiency with a primary language other than Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain | Up to 30 minutes
  Participants will be asked to rate their pain on a visual analog pain scale. The scale is rated from 0 (no pain) to 10 (pain as bad as it can be)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Formica, DDS, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No